CLINICAL TRIAL: NCT06949046
Title: Effects of a Nursing-led Communication Support Program Using Mobile Health Information on Physical and Mental Status in Breast Cancer Patients Undergoing Concurrent Chemotherapy: a Randomized Controlled Trial
Brief Title: Effects of a Nursing-led Communication Using Mobile Health Information in Breast Cancer Patients Undergoing Concurrent Chemotherapy
Acronym: breast cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Mei Man, Student, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: A202405082; A202405082 (Registry Identifier: Tri-Service General Hospital Institutional Review Board)
Record Dates: First submitted 2024-10-04; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: breast cancer; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nursing-led communication (Experimental): nursing-led communication support
  Interventions: Other: nursing-led communication support
- Nursing routine treatment (Placebo Comparator): Nursing routine treatment
  Interventions: Other: Nursing routine treatment

INTERVENTIONS:
Other: nursing-led communication support — nursing-led communication support program using mobile health information
  Arms: nursing-led communication
Other: Nursing routine treatment — Nursing routine treatment
  Arms: Nursing routine treatment

SUMMARY:
Breast cancer is the most common malignant tumor among women. Side effects from initial chemotherapy include sleep disorders, anxiety, depression, and reduced quality of life. Mental health distress is also a major issue in cancer care. This study integrates mobile health information with a nurse-led communication support plan, aiming to improve patients' physical and mental outcomes during chemotherapy.

DETAILED DESCRIPTION:
The objective of this study is to explore the effects of a nursing-led communication support program using mobile health information on physical and mental state in breast cancer patients undergoing initial chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

breast cancer initial chemotherapy

Exclusion Criteria:

Patients whose cancer has recurred without undergoing the first course of chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Effects of a nursing-led communication support program using mobile health information on physical and mental status in breast cancer patients undergoing concurrent chemotherapy: a randomized controlled trial | 1 year
  Used the Quality of life questionnaire test

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No